CLINICAL TRIAL: NCT04567446
Title: Discovery of Microbiome-based Biomarkers for Patients With Cancer Using Metagenomic
Brief Title: Discovery of Microbiome-based Biomarkers for Patients With Cancer Using Metagenomic Approach
Acronym: ONCOBIOTICS
Status: Recruiting | Type: Observational
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A02010-53; 2017/2619 (Other: CSET number)
Record Dates: First submitted 2020-02-10; First posted 2020-09-28 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Defecation; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with bladder cancer who will start cancer treatment: Collection of biological samples (stool and blood) and data from patients included in the study will be performed:
  1. By identifying the patients who will start treatment anticancer (chemotherapy, hormone therapy, immunotherapy).
  2. Collection of biological resources (all samples will be collected in fresh): stool and blood
  3. Collection of clinical data corresponding to each patient included in the study by a clinical research assistant
  Interventions: Other: Stool; Other: Blood sample
- Patients with Non-Small-Cell Lung cancer who will start cancer treatment: Collection of biological samples (stool and blood) and data from patients included in the study will be performed:
  1. By identifying the patients who will start treatment anticancer (chemotherapy, hormone therapy, immunotherapy).
  2. Collection of biological resources (all samples will be collected in fresh): stool and blood
  3. Collection of clinical data corresponding to each patient included in the study by a clinical research assistant
  Interventions: Other: Stool; Other: Blood sample
- Patients with kidney cancer who will start cancer treatment: Collection of biological samples (stool and blood) and data from patients included in the study will be performed:
  1. By identifying the patients who will start treatment anticancer (chemotherapy, hormone therapy, immunotherapy).
  2. Collection of biological resources (all samples will be collected in fresh): stool and blood
  3. Collection of clinical data corresponding to each patient included in the study by a clinical research assistant
  Interventions: Other: Stool; Other: Blood sample

INTERVENTIONS:
Other: Stool — collection at baseline (or before the third injection), at the first evaluation (CT-scan), at ≥ 6 months after the first injection, at toxicity and at relapse, at 1 week after the end of antibiotics treatment
Other: Blood sample — 20 mL collection at baseline (or before the third injection), at the first evaluation (CT-scan), at ≥ 6 months after the first injection, at toxicity and at relapse, at 1 week after the end of antibiotics treatment

SUMMARY:
Multicentric prospective study with collection of biological samples as part of type II research

ELIGIBILITY:
Inclusion Criteria:

* Patient with cancer who will start treatment anticancer (see cohorts).
* Patient information and signature of the consent form before any specific procedure for the study. The patient must be able and must be inclined to cooperate in the study procedures.
* Patient affiliated to a social security scheme or beneficiary of a similar scheme.

Exclusion Criteria:

* Pregnant or lactating woman
* Patient under guardianship or curatorship or deprived of liberty by a decision judicial or administrative or patient unable to give his consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with cancer who will start treatment anticancer
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 2 years
  To define metagenomic signatures associated with cancer

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Gustave Roussy, Villejuif, Val De Marne
  - Centre hospitalier du Pays d'Aix, Aix-en-Provence
  - Centre Pierre Curie, Beuvry
  - Clinique du Flandre, Coudekerque-Branche
  - CHRU Lille - Hôpital Calmette, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital St Louis, Paris
  - Hôpital Foch, Suresnes
  - Centre hospitalier TOULON - Sainte-Musse, Toulon

IPD SHARING:
Plan to Share IPD: Undecided